CLINICAL TRIAL: NCT02899572
Title: Impact of a Sexology Consultation on Diabetes Disease Control of Type 2 Male Diabetics With Erectile Dysfunction: a Monocentric Randomised Comparative Study
Brief Title: Impact of a Sexology Consultation on Disease Control of Type 2 Male Diabetics With Erectile Dysfunction
Acronym: RADOTES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/CHU/01
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Erectile Dysfunction; Type 2 Diabetes
MeSH Terms: conditions — Erectile Dysfunction; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sexology consultation (Experimental): specialized sexology consultation planned in the 15 days after inclusion. Randomisation is performed at D7 during a phone call to the patient.
  Interventions: Procedure: Sexology consultation
- Leaflet concerning erectile disorders (No Intervention): leaflet explaining erectile disorders related to type 2 diabetes will be sent by post to the patients. Randomisation is performed at D7 during a phone call to the patient.

INTERVENTIONS:
Procedure: Sexology consultation — a sexology consultation is planned in the 15 days after inclusion
  Arms: Sexology consultation

SUMMARY:
Erection disorders constitute the first sign of vascular injury in type 2 diabetes patients. The important frequency of these disorders and their consequences in term of quality of life have a strong contrast with the actual interest showed for them by the medical community.

Natural evolution of the disease and its management make that these disorders often occur little time after a therapeutic change. As a consequence, patients often accuse their medication to be responsible for the appearance of these disorders. This confusion, associated to false believes that may have the patients on their disease or their treatment, often leads to treatment discontinuation which has a deleterious effect on the disease evolution.

Educational therapy programs showed a positive impact on therapeutic adherence. Increasing patients' knowledge on their disease and treatments increases their therapeutic adherence and makes it easier to balance diabetes and therefore limits complications appearance.

Educational therapy programs concern today the disease, its process, its evolution, its treatments, their efficacy, their adverse effects but erection disorders are not specifically addressed.

This study aims to evaluate the impact of a sexology consultation on diabetes balance measured via HbA1c rate. This consultation aims at precising this particular symptom of erection disorders, without any medicine prescription. The aim is to explain to patients the different links between their symptoms, diabetes, medicines and themselves.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic male medically treated
* aged from 18 to 65 years old included
* having issue obtaining or maintaining an erection allowing a satisfying sexual intercourse
* hospitalised or followed in consultation in one of the 2 participating sites

Exclusion Criteria:

* treated by a medicine which could be responsible for the erectile disorders (beta-blockers, central anti-hypertensive drugs, antialdosterones)
* presenting another disease which could be responsible for the erectile disorders (neurological, hormonal, vascular, psychiatric diseases)
* treated by an insulin pump

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-10 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of HbA1c according to the randomisation group | 3 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Céline REGNIER, MD, Principal Investigator — CH Gabriel Martin
Locations (1):
- Centre Hospitalier Gabriel Martin, Saint-Paul, France

IPD SHARING:
Plan to Share IPD: No